CLINICAL TRIAL: NCT06418672
Title: Go Sun Smart Georgia Evaluation
Acronym: GSSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Klein Buendel, Inc. (Industry)
Responsible Party: Principal Investigator, Alexandra Morshed, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00007062; 3U48DP006377-03S4 (NIH)
Record Dates: First submitted 2024-05-01; First posted 2024-05-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Sun Safety
Keywords: Sun Protection Behavior; Sun Safety Education

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Intervention (Experimental): 6 worksites will be enrolled. GSSG implementation in May-August 2024
  Interventions: Behavioral: Go Sun Smart Georgia (GSSG)
- Delayed Intervention (Active Comparator): 6 worksites will be enrolled. GSSG implementation in August- December 2024.
  Interventions: Behavioral: Go Sun Smart Georgia (GSSG)

INTERVENTIONS:
Behavioral: Go Sun Smart Georgia (GSSG) — Go Sun Smart Georgia (GSSG) is an educational, train-the-trainer, and technical assistance program for Georgia worksites that employ outdoor workers.
  GSSG is delivered through personal contacts with senior worksite managers, employee training, and distribution of educational materials. In meetings with managers, trained coaches work to increase perceived need for workplace sun safety, cite advice from national authorities (e.g., CDC and NIOSH), plan for policy implementation, alter policies/education and/or workplace to improve fit, clarify changes to other managers/ employees, and bundle sun safety with worksite safety.
  The intervention period will last 12-16 weeks in each of the groups.

SUMMARY:
The goal of this clinical trial is to evaluate the dissemination of the Go Sun Smart Georgia (GSSG) program with Georgia worksites and learn whether the intervention changes the employees' sun protection behavior in outdoor workers in Southwest Georgia.

The primary aim is to assess program effectiveness by comparing employee sun protection practices between the employers assigned to the GSSG intervention and the employers assigned to the wait-list control group (delayed intervention). The hypothesis that will be tested is that compared to the delayed intervention group, employees at intervention worksites will practice more sun protection during the post-test.

Worksites will be asked to complete internal coach training and participate in technical assistance around sun safety. Study participants will fill out surveys and participate in interviews

DETAILED DESCRIPTION:
This project builds on the original Go Sun Smart at Work (GSSW) program-a sun safety educational program delivered to worksite leaders, managers, and workers-that was previously shown to be effective for employers adopting sun safety policies and implementing sun safety education and actions, and improved employees' sun protection behavior (e.g., use of protective clothing).

To successfully implement and scale up GSSW with outdoor workers in Southwest Georgia-predominantly African American and Hispanic-this intervention must be systematically adapted to ensure program fit to the population and setting while maintaining core program elements. A well-adapted and tailored occupational sun safety program with high dissemination potential will greatly impact this overlooked employee population, reduce health care costs, improve quality of life, and save lives. The adaptation process took place in 2022-2024, and the adapted Go Sun Smart Georgia (GSSG) program will be evaluated in 2024.

Go Sun Smart Georgia (GSSG) is an educational, train-the-trainer, and technical assistance program for Georgia worksites that employ outdoor workers. It will be implemented with worksites assigned to the intervention group in May-Aug 2024 and with worksites assigned to the comparison (delayed intervention) group in Aug - Dec. 2024. The study team will provide worksites with training for internal worksite coaches (the coach(es) will be employee(s) chosen by the worksite to serve as a champion for the program, not part of the study staff and paid by the worksite), training for other internal educators, technical assistance for conducting the program, and employee educational sessions, as needed.

ELIGIBILITY:
Inclusion Criteria:

Outdoor workers

* Employed at participating worksite
* Works at least 5 hours outdoors per week
* Can read and/or clearly understand English

Managers

* Employed at participating worksite in supervisory position
* Responsible for worksite safety/health policy or training
* Can read and/or clearly understand English

Semi-structured interviews

* Employed by participating worksite
* Closely involved with GSSG implementation
* Can read and/or clearly understand English

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Cognitively impaired or Individuals with Impaired Decision-Making Capacity
* Individuals who are not able to clearly understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in outdoor worker sun safety behaviors | 16 weeks
  Will be captured through outdoor worker survey (posttest). To evaluate the impact of GSSG on sun safety behaviors (primary outcome), employees will report a) frequency of sun protection at work (i.e., sunscreen with SPF 30+, long-sleeved shirts, long pants, hat with wide-brim, sunglasses, shade use, limit midday sun exposure, and have sunscreen, hat and eye protection at all times [1=never, 5=always]) and b) sunburn in past 3 months on the job (yes/no; number).
  Surveys will include questions about amount of times respondent works outdoors; the respondent's sun and heat protection behaviors; perceptions of their sun exposure risk and history of sunburn; presence and perception of workplace policies, procedures, standards, resources, and training for sun safety and heat at the organization; experience with the Go Sun Smart Georgia program; and respondent demographics.

SECONDARY OUTCOMES:
Change in worksite policy adoption | Baseline, After 16 weeks
  Will be captured through manager survey, outdoor worker survey
Worksite sun safety education | Baseline, After 16 weeks
  Will be captured through manager survey, outdoor worker survey
Change in worksite sun safety actions | Baseline, After 16 weeks
  Will be captured through manager survey
Appropriateness of program | At 16 weeks
  Will be captured through manager survey, outdoor worker survey, semi-structured interviews
Feasibility of program | At 16 weeks
  Will be captured through manager survey, outdoor worker survey, semi-structured interviews
Acceptability of program | At 16 weeks
  Will be captured through manager survey, outdoor worker survey, semi-structured interviews
Fidelity of implementation | 16 weeks
  Will be captured through program logs.
Representativeness of participants | At 16 weeks
  Will be captured through outdoor worker survey

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Morshed, PhD, Principal Investigator — Rollins School of Public Health
Locations (1):
- Rollins School of Public Health, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
To enable interoperability of datasets and resources, we will provide a data codebook/dictionary for all variables included per dataset and documentation with the following elements: information about how the data were collected, sampling details, data cleaning details, related publications, and grant information. The team will make available platform-independent, character-based formats of datasets (e.g., CSV) that retain full detail and precision
Supporting Information: SAP, CSR
Time Frame: Data will be made available no later than the time of an associated publication or the end of the performance period of the SIP award that funds this project. Data will be made available for at least 5 years.
Access Criteria: Scientific data will be preserved and shared using the Emory Dataverse Repository, sco.library.emory.edu/dataverse, where they will be publicly available to those interested in using them.